CLINICAL TRIAL: NCT00231816
Title: A Double-Blind, Randomized, Multicenter Study to Evaluate the Safety, Tolerability, and Immunogenicity of V211 Administered Concomitantly Versus Nonconcomitantly With Influenza Virus Vaccine (Inactivated)
Brief Title: A Study of an Investigational Zoster Vaccine in Subjects With a History of Varicella (Chickenpox) Given Concomitantly With Another Vaccine (V211-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-011; 2005_036
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Herpes Zoster
Keywords: Prevention of Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine; Influenza Vaccines; vaxigrip

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Concomitant (Experimental): Zostavax concomitantly with influenza vaccine on Day 1, placebo at week 4
  Interventions: Biological: ZOSTAVAX™ (concomitant); Biological: Comparator: Influenza Vaccine
- Nonconcomitant (Experimental): Influenza vaccine and Zostavax placebo on Day 1, Zostavax at week 4
  Interventions: Biological: Comparator: Influenza Vaccine; Biological: ZOSTAVAX™ (Nonconcomitant)

INTERVENTIONS:
Biological: ZOSTAVAX™ (concomitant) — a single administration of 0.65 mL subcutaneous injection of zoster vaccine live on Day 1 and placebo at Week 4
  Other Names: V211
  Arms: Concomitant
Biological: Comparator: Influenza Vaccine — a single administration of 0.5 mL intramuscular injection of influenza vaccine (inactivated) at Day 1
  Other Names: Fluzone, Vaxigrip
Biological: ZOSTAVAX™ (Nonconcomitant) — Placebo injection on Day 1 and a single administration of 0.65 mL subcutaneous injection of zoster vaccine live at Week 4
  Arms: Nonconcomitant

SUMMARY:
The purpose of this study is to determine whether the investigational zoster vaccine has a comparable immune response (the body's ability to protect against disease) and safety profile when given concomitantly with another vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Adults 50 years of age or older

Exclusion Criteria:

* Prior history of Herpes Zoster (shingles)
* Prior receipt of varicella or zoster vaccine
* Immunosuppressed

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 2005-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Kerzner B, Murray AV, Cheng E, Ifle R, Harvey PR, Tomlinson M, Barben JL, Rarrick K, Stek JE, Chung MO, Schodel FP, Wang WW, Xu J, Chan IS, Silber JL, Schlienger K. Safety and immunogenicity profile of the concomitant administration of ZOSTAVAX and inactivated influenza vaccine in adults aged 50 and older. J Am Geriatr Soc. 2007 Oct;55(10):1499-507. doi: 10.1111/j.1532-5415.2007.01397.x. PMID 17908055
- [Background] Sutradhar SC, Wang WW, Schlienger K, Stek JE, Xu J, Chan IS, Silber JL. Comparison of the levels of immunogenicity and safety of Zostavax in adults 50 to 59 years old and in adults 60 years old or older. Clin Vaccine Immunol. 2009 May;16(5):646-52. doi: 10.1128/CVI.00407-08. Epub 2009 Mar 4. PMID 19261769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 13 sites in the United States and 7 sites in Europe.
  First Patient In (FPI): 23-SEP-2005; Last Patient Last Visit (LPLV): 08-MAR-2006
Groups:
- Concomitant Group: ZOSTAVAX™ 0.65 mL subcutaneous (SC) injection administered concomitantly with 0.5 mL intramuscular (IM) influenza vaccine injection at separate injection sites on Day 1 and placebo injection at Week 4
- Nonconcomitant Group: Influenza vaccine 0.5 mL IM injection administerd with placebo injection on Day 1 and ZOSTAVAX™ 0.65 mL SC injection at Week 4
Period: Overall Study
Arm/Group | Concomitant Group | Nonconcomitant Group
Started | 382 | 381
Vaccinated at Visit 1 | 382 | 380 (One participant was randomized but not vaccinated)
Vaccinated at Visit 2 | 369 | 371
Completed | 366 (Participant received required vaccines and returned completed vaccination report cards at Visits 2&3) | 369 (Participant received required vaccines and returned completed vaccination report cards at Visits 2&3)
Not Completed | 16 | 12
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 8 | 5
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Group | Nonconcomitant Group | Total
Number analyzed (Participants) | 382 | 380 | 762
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.99) | 63.6 (8.24) | 63.5 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 212 | 427
  Male | 167 | 168 | 335
Race/Ethnicity, Customized [Number; unit: participants]
  African | 1 | 0 | 1
  Asian | 5 | 4 | 9
  Black | 106 | 100 | 206
  Hispanic American | 11 | 11 | 22
  Indian | 0 | 1 | 1
  Multiracial | 0 | 2 | 2
  Native American | 1 | 1 | 2
  White | 258 | 261 | 519

OUTCOME MEASURES:

1. Primary Outcome: Varicella-zoster Virus (VZV) Glycoprotein Enzyme-linked Immunosorbent Assay (gpELISA) Antibody Responses
Description: The Geometric mean titer (GMT) of the VZV glycoprotein enzyme-linked immunosorbent assay (gpELISA) antibody responses at Week 4 postvaccination in participants who received ZOSTAVAX™ concomitantly with influenza vaccine was compared to that in subjects who received influenza vaccine and ZOSTAVAX™ nonconcomitantly.
Time Frame: 4 weeks
Population: The primary analysis was based on the per protocol population defined as participants who had valid GMT results from samples obtained within the prespecified day ranges at Day 1, at Week 4, or at Week 8 postvaccination, and who did not meet any of the protocol violations prespecified in the statistical analysis plan (SAP).
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Concomitant Group | Nonconcomitant Group
Number analyzed (Participants) | 361 | 366
gpELISA units/mL | 553.5 [499.0 to 613.9] | 588.7 [531.9 to 651.5]

2. Other Pre Specified Outcome: Geometric Mean Fold Rise (GMFR) in VZV gpELISA Antibody Titers From Prevaccination to 4 Weeks Postvaccination
Description: GMFR of the VZV gpELISA antibody titers from prevaccination
  to 4 weeks postvaccination when ZOSTAVAX™ is administered concomitantly with influenza vaccine
Time Frame: prevaccination to 4 weeks postvaccination
Population: The analysis was based on the per protocol population defined as participants who had valid GMFR results from samples obtained within the prespecified day ranges at Day 1, at Week 4, or at Week 8 postvaccination, and who did not meet any of the protocol violations prespecified in the statistical analysis plan (SAP)
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Groups:
- Concomitant Group: ZOSTAVAX™ 0.65 mL SC injection administered comcomitantly with 0.5 mL IM influenza vaccine injection at separate injection sites on Day 1 and placebo injection at Week 4
Arm/Group | Concomitant Group
Number analyzed (Participants) | 354
ratio | 2.1 [2.0 to 2.3]

3. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of H1N1 Strain Antibody Responses at 4 Weeks Postvaccination
Description: GMT of the H1N1 strain antibody responses at 4 weeks postvaccination in participants who receive ZOSTAVAX™ concomitantly with influenza vaccine and those who receive ZOSTAVAX™ and influenza vaccine nonconcomitantly
Time Frame: 4 weeks postvaccination
Population: The analysis was based on the per protocol population defined as participants who had valid results from samples obtained within the prespecified day ranges at Day 1, at Week 4, or at Week 8 postvaccination, and who did not meet any of the protocol violations prespecified in the SAP.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Concomitant Group | Nonconcomitant Group
Number analyzed (Participants) | 363 | 363
titers | 122.9 [107.8 to 140.0] | 134.2 [118.3 to 152.2]

4. Other Pre Specified Outcome: GMTs of H3N2 Strain Antibody Responses at 4 Weeks Postvaccination
Description: GMT of the H3N2 strain antibody responses at 4 weeks postvaccination in participants who receive ZOSTAVAX™ concomitantly with influenza vaccine and those who receive ZOSTAVAX™ and influenza vaccine nonconcomitantly
Time Frame: 4 weeks postvaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Concomitant Group | Nonconcomitant Group
Number analyzed (Participants) | 363 | 363
titers | 162.7 [140.4 to 188.4] | 150.5 [129.8 to 174.5]

5. Other Pre Specified Outcome: GMTs of B Strain Antibody Responses at 4 Weeks Postvaccination
Description: GMT of the B strain antibody responses at 4 weeks postvaccination in participants who receive ZOSTAVAX™ concomitantly with influenza vaccine and those who receive ZOSTAVAX™ and influenza vaccine nonconcomitantly
Time Frame: 4 weeks postvaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Concomitant Group | Nonconcomitant Group
Number analyzed (Participants) | 363 | 363
titers | 119.8 [104.8 to 137.1] | 136.5 [120.5 to 154.7]

ADVERSE EVENTS:
Time Frame: Day 1-28 following each vaccination
Description: Injection-site adverse events (AEs), rashes, oral temperatures (if the subject felt febrile), and other AEs were recorded by the participant on a Vaccination Report Card which was reviewed by the study site personnel at the end of each 28-day follow-up period.
  4 participants from each group were lost to follow up & not included in the analysis
Arm/Group | Concomitant Group | Nonconcomitant Group
Serious Adverse Events (participants affected / at risk) | 6/378 | 5/376
Other Adverse Events (participants affected / at risk) | 199/378 | 181/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant Group (N=378) | Nonconcomitant Group (N=376)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant Group (N=378) | Nonconcomitant Group (N=376)
Upper respiratory tract infection (Infections and infestations) | 19 | 17
Injection Site Erythema (Influenza vaccine injection site) (General disorders) | 46 | 29
Injection Site Erythema (Placebo injection site) (General disorders) | 11 | 19
Injection Site Erythema (ZOSTAVAX™ injection site) (General disorders) | 125 | 101
Injection Site Pain (Influenza vaccine injection site) (General disorders) | 90 | 86
Injection Site Pain (Placebo injection site) (General disorders) | 16 | 23
Injection Site Pain (ZOSTAVAX™ injection site) (General disorders) | 114 | 107
Injection Site Swelling (Influenza vaccine injection site) (General disorders) | 41 | 31
Injection Site Swelling (ZOSTAVAX™ injection site) (General disorders) | 70 | 94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.